CLINICAL TRIAL: NCT07266025
Title: Adebrelimab Combined With Induction Chemotherapy or SHR-8068 for Mismatch Repair-Deficient/Microsatellite Instability-High (dMMR/MSI-H) Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma：A Randomized, Non-comparative Phase 2 Study
Acronym: CATALIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuefei.Wang, Chief of Department of Gastrointestinal Surgery, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025379
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Adenocarcinoma; Mismatch Repair Deficient or MSI-High Solid Tumors; Immunotherapy
MeSH Terms: conditions — Turcot syndrome | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants assigned to arm 1 will receive neoadjuvant adebrelimab 1200 mg intravenously on day 1 combined with XELOX (capecitabine 1000 mg/m² orally twice daily on days 1-14 plus oxaliplatin 130 mg/m² intravenously on day 1) for one cycle, followed by adebrelimab monotherapy at the same dose and schedule for three additional cycles. Within 4-6 weeks after completion of the fourth cycle, curative-intent D2 radical gastrectomy will be performed. Post-operative adjuvant systemic therapy-regimen, duration, and number of cycles-will be left to the discretion of the treating investigator, guided by institutional standards and the patient's pathological and clinical status.
  Interventions: Drug: Adebrelimab; Drug: XELOX; Procedure: D2 radical gastrectomy
- Arm 2 (Experimental): Participants in arm 2 will receive neoadjuvant adebrelimab 1200 mg plus SHR-8068 280 mg administered intravenously on day 1 of a 21-day cycle for one cycle, followed by adebrelimab 1200 mg monotherapy on day 1 every 3 weeks for three additional cycles. Curative-intent D2 radical gastrectomy is scheduled 4-6 weeks after completion of the fourth cycle. Any post-operative adjuvant systemic treatment-including regimen, duration, and number of cycles-will be determined at the investigator's discretion according to institutional guidelines and the patient's pathological and clinical status.
  Interventions: Drug: Adebrelimab; Drug: SHR-8068; Procedure: D2 radical gastrectomy

INTERVENTIONS:
Drug: Adebrelimab — Participants in both arms will receive neoadjuvant adebrelimab 1200mg intravenously on day 1 of a 21-day cycle for four cycles.
Drug: XELOX — Participants assigned to arm 1 will receive neoadjuvant XELOX (capecitabine 1000 mg/m² orally twice daily on days 1-14 plus oxaliplatin 130 mg/m² intravenously on day 1) for one cycle.
  Arms: Arm 1
Drug: SHR-8068 — Participants assigned to arm 2 will receive SHR-8068 280 mg administered intravenously on day 1 for one cycle.
  Arms: Arm 2
Procedure: D2 radical gastrectomy — Curative-intent D2 radical gastrectomy is scheduled 4-6 weeks after completion of the fourth cycle.

SUMMARY:
This is a randomized, non-comparative, open-label, two-arm phase II clinical trial designed to evaluate the efficacy and safety of neoadjuvant therapy with adebrelimab plus induction chemotherapy versus adebrelimab plus SHR-8086 in patients with dMMR/MSI-H gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years
* Pathologically confirmed gastric or gastro-oesophageal-junction adenocarcinoma (Siewert II and III only)
* dMMR confirmed by IHC or MSI-H confirmed by PCR
* Investigator-assessed potentially curative resection feasible before study entry
* CT or MRI clinical stage cT ≥ 2 N any M0 per AJCC 8th edition; laparoscopy with peritoneal washing cytology (and peritoneal biopsy if indicated) recommended to exclude peritoneal metastasis
* ECOG performance status 0-2
* Able to swallow tablets
* Expected survival ≥ 6 months
* Laboratory values within 7 days before randomisation:

ANC > 1.5 × 10⁹/L, Hb ≥ 80 g/L, PLT ≥ 75 × 10⁹/L Serum creatinine ≤ 1.5 × ULN or eGFR ≥ 60 mL/min/1.73 m² ALT and AST ≤ 2.5 × ULN; total bilirubin ≤ 1.5 × ULN (or TBIL > 1.5 × ULN with direct bilirubin ≤ ULN); albumin ≥ 25 g/L INR or PT ≤ 1.5 × ULN and aPTT ≤ 1.5 × ULN (or on anticoagulation within therapeutic range)

* Signed written informed consent; able to comply with protocol visits, treatment, labs, biospecimen collection
* WOCBP must have negative serum pregnancy test within 72 h before randomisation, not breastfeeding, and use highly effective contraception from screening until 2 months after last adebrelimab/SHR-8068 or 6 months after last chemotherapy, whichever is longer
* Men with pregnant partners or WOCBP partners must be surgically sterile or use highly effective contraception during study and for same post-treatment periods; no sperm donation allowed

Exclusion Criteria:

* Tumour histology squamous-cell, neuro-endocrine, or other non-adenocarcinoma types
* Unresectable disease (tumour-related or surgical contraindication) or subject refuses surgery
* Tumour requiring transthoracic surgical approach
* CNS metastases and/or carcinomatous meningitis
* Prior anti-gastric-cancer therapy (surgery, radiotherapy, chemotherapy, targeted, immunotherapy) except bypass for obstruction
* Previous malignancy or concurrent malignancy except completely excised basal/squamous skin cancer, superficial bladder cancer, or in-situ prostate/cervix/breast cancer disease-free ≥ 5 years
* Cardiac conditions:

NYHA class > II or LVEF < 50 % on echo Unstable angina MI within 1 year Resting QTc > 450 ms (M) or > 470 ms (F) Clinically significant ECG abnormalities, complete LBBB, 3rd-degree AV block, 2nd-degree AV block, PR > 250 ms Risk factors for QT prolongation (HF, hypokalaemia, congenital long-QT syndrome, family history of long QT or sudden death < 40 y, concomitant QT-prolonging drugs)

* History of GI perforation, intra-abdominal abscess, or bowel obstruction within 3 months or imaging/clinical signs of obstruction
* Clinically significant bleeding or bleeding diathesis within 3 months (e.g. GI bleeding, haemorrhagic gastritis, vasculitis); positive faecal occult blood must be endoscopically cleared if still positive on repeat testing (unless gastroscopy within 3 months shows no lesion)
* Arterial or venous thrombo-embolic event within 6 months (stroke, TIA, intracranial haemorrhage, cerebral infarction)
* Hypersensitivity to any study-drug component
* Severe hypersensitivity history to any monoclonal antibody
* Pregnant or lactating women
* Positive HIV antibody
* Active hepatitis (HBsAg positive with HBV DNA ≥ 500 IU/mL; HCV antibody positive with HCV RNA > ULN)
* Prior therapy targeting CTLA-4/PD-1/PD-L1 or other T-cell co-stimulatory/immune-checkpoint pathways (including therapeutic vaccines)
* Active autoimmune disease or autoimmune disease with relapse risk within 2 years (except stable hypothyroidism on replacement or well-controlled type 1 diabetes on insulin)
* History of idiopathic pulmonary fibrosis, drug-related pneumonia, organising pneumonia (BOOP/COP), or CT evidence of active pneumonia at screening
* Live attenuated vaccine within 4 weeks before first study dose or expected need during study
* Immunodeficiency disorder or chronic systemic corticosteroids or other immunosuppressive therapy within 7 days before first dose (includes prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-TNF agents)
* Any condition that, in the investigator's opinion, increases study risk, interferes with protocol conduct, or compromises informed consent or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | From randomization to the date of surgery, an average of 14 weeks.
  The proportion of participants in whom no viable tumor cells remain in the primary tumor bed and regional lymph nodes (ypT0N0).

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | From randomization to the date of surgery, an average of 14 weeks.
  The proportion of participants in whom residual viable tumor cells constitute <10 % of the primary tumor bed in the resected surgical specimen.
ypN stage | From randomization to the date of surgery, an average of 14 weeks.
  Lymph-node status after neoadjuvant therapy (ypN stage) will be assessed according to the American Joint Committee on Cancer (AJCC) 8th edition staging system.
R0 resection rate | From randomization to the date of surgery, an average of 14 weeks.
  The proportion of patients who undergo surgery with microscopically negative resection margins.
Event-free survival (EFS) | The time from randomization to documented disease progression, disease recurrence, or death from any cause, whichever occurs first, assessed up to 5 years.
Overall survival (OS) | The time from randomization to death from any cause, assessed up to 5 years.

IPD SHARING:
Plan to Share IPD: No